CLINICAL TRIAL: NCT04166942
Title: A Single-dose, Open-label, Pharmacokinetic Study of KD025 in Subjects With Normal Hepatic Function & Subjects With Varying Degrees of Hepatic Impairment
Brief Title: KD025 Hepatic Impairment Study With Normal Hepatic Function and Subjects With Varying Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP17629; KD025-109 (Other: Kadmon)
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — KD025; belumosudil

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, parallel-group study with the following subject treatment arms:
  Group 1: normal hepatic function; Group 2: mild hepatic impairment; Group 3: moderate hepatic impairment; Group 4: severe hepatic impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Group 1--Control) (Experimental): Matched healthy subjects with normal hepatic function
  Interventions: Drug: KD025
- Mild Hepatic Impairment (Group 2) (Experimental): Subjects with mild hepatic impairment based on Child-Pugh Class A score of 5 or 6
  Interventions: Drug: KD025
- Moderate Hepatic Impairment (Group 3) (Experimental): Subjects with moderate hepatic impairment based on Child-Pugh Class B score of 7 to 9
  Interventions: Drug: KD025
- Severe Hepatic Impairment (Group 4) (Experimental): Subjects with severe hepatic impairment based on Child-Pugh Class C score of 10 to 14
  Interventions: Drug: KD025

INTERVENTIONS:
Drug: KD025 — Single dose of 200 mg KD025 orally
  Other Names: belumosudil

SUMMARY:
This is a study to characterize the pharmacokinetics, safety and tolerability of KD025 and KD025 metabolites in subjects with mild, moderate or severe hepatic impairment compared to healthy subjects with normal hepatic function.

DETAILED DESCRIPTION:
The primary objective of the study is:

• To assess the pharmacokinetics (PK) of KD025 following a single oral dose of KD025 in subjects with mild, moderate, or severe hepatic impairment compared to healthy subjects with normal hepatic function.

The secondary objectives of the study are:

* To evaluate the safety and tolerability of a single oral dose of KD025 in subjects with mild, moderate, or severe hepatic impairment, and in healthy subjects with normal hepatic function.
* To assess the PK of the KD025 metabolites following a single oral dose of KD025 in subjects with mild, moderate, or severe hepatic impairment compared to healthy subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

For All Subjects:

Subjects must satisfy all of the following criteria at the Screening visit, unless otherwise stated:

1. Males or females, of any race, between 18 and 75 years of age, inclusive.
2. Body mass index between 18.0 and 38.0 kg/m^2, inclusive.
3. Females of non-childbearing potential defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal (defined as females at least 45 years of age with at least 12 months post-cessation of menses without an alternative medical cause, even with a follicle-stimulating hormone level ≤40 mIU/mL, unless on hormone replacement therapy).
4. Males will agree to use contraception
5. Male subjects must not donate sperm from Check-in (Day -1) until 90 days after the Follow-up visit.
6. Able to comprehend and willing to sign an informed consent form and to abide by the study restrictions.

   For Subjects with Normal Hepatic Function Only:
7. In good health, determined by no clinically significant findings from medical history, PE, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and Check-in (Day -1), as assessed by the Investigator (or designee).
8. Matched to subjects with mild, moderate, or severe hepatic impairment in sex, age (±10 years), and body mass index (±20%).

   For Subjects with Hepatic Impairment Only:
9. Documented chronic stable liver disease (Child-Pugh Class A [mild], B [moderate], or C [severe] at Screening); diagnosis of hepatic impairment due to parenchymal liver disease. If the Child-Pugh Class of a subject differs between Screening and Check-in, the Child-Pugh Class documented at Screening will be utilized for enrollment. This will exclude biliary liver cirrhosis or other causes of hepatic impairment unrelated to parenchymal disorder.:

   * 'Documented' is defined by at least 1 of the following: medical history, PE, hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging, and/or liver biopsy.
   * 'Chronic' is defined as >6 months.
   * 'Stable' is defined as no clinically significant change in disease status within the last 3 months (90 days), as documented by the subject's recent medical history (eg, no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time by more than 50%).
10. Subjects with mild, moderate, or severe hepatic impairment may have medical findings consistent with their hepatic dysfunction as determined by medical history, PE, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and Check-in (Day -1), as assessed by the Investigator (or designee).
11. Non-hepatic, abnormal clinical laboratory evaluations not clinically relevant, as judged by the Investigator (or designee) and Covance Medical Monitor.
12. Currently on a stable medication regimen, defined as not starting new drug(s) or changing drug dose(s) within 30 days of administration of study drug (Day 1). Concomitant medications administered within 30 days prior to administration of KD025 (Day 1) must be approved by the Investigator (or designee), Sponsor, and Covance Medical Monitor.
13. Anemia secondary to hepatic disease will be acceptable, if hemoglobin >9 g/dL and anemia symptoms are not clinically significant as judged by the Investigator (or designee) and Covance Medical Monitor.
14. Platelet count ≥35 × 10^9 platelets/L.
15. Subjects with diabetes mellitus may be included, provided the subjects have:

    1. Glycosylated hemoglobin A1c values ≤9.5% at Screening. Subjects with values outside this range may be allowed by the Covance Medical Monitor on a case-by-case basis.
    2. Blood glucose values ≤240 mg/dL at Screening and Check-in (Day -1) while on subjects' normal diabetes medication.

Exclusion Criteria:

Subjects will be excluded from the study if they satisfy any of the following criteria at the Screening visit, unless otherwise stated:

For All Subjects:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Clinically significant physical examination abnormality, as determined by the Investigator (or designee).
5. Use or intend to use any drugs known to be moderate or strong inhibitors or inducers of CYP3A4 within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee) in consultation with the Covance Medical Monitor.
6. Use or intend to use any proton pump inhibitors or H2 antagonists within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee) in consultation with the Covance Medical Monitor.
7. Use or intend to use any phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee).
8. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
9. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
10. Positive urine drug screen at Screening and/or Check-in (Day -1) that is not otherwise explained by permitted concomitant medication, or positive alcohol test result at Check-in (Day -1). Either a breath or urine alcohol test may be performed in accordance with the standard practice of each CRU.
11. Positive human immunodeficiency virus test.
12. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (whichever is longer) of the investigational drug, prior to dosing.
13. Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to Check-in (Day -1).
14. Receipt of blood products within 2 months prior to Check-in.
15. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
16. Poor peripheral venous access.
17. Have previously completed or withdrawn from this study or any other study investigating KD025, and have previously received KD025.
18. Subjects who, in the opinion of the Investigator (or designee) should not participate in this study.

    For Subjects with Normal Hepatic Function Only:
19. QT interval corrected for heart rate using Fridericia's method (QTcF) >450 ms confirmed by repeat measurement.
20. Evidence of hepatorenal syndrome and/or estimated creatinine clearance range <90 mL/min, as determined by the Investigator (or designee), calculated using the Cockcroft-Gault equation at Screening and Check-in (Day -1).

    For male subjects: ([1.23 × {140-age} × {weight in kg})])/(serum creatinine in μmol/L) For female subjects: ([1.04 × {140-age} × {weight in kg})])/(serum creatinine in μmol/L)
21. Ventricular dysfunction or history of risk factors for Torsade de Pointes (e.g., unexplained syncope, known long QT syndrome, heart failure, and cardiomyopathy). Subjects will be excluded if there is a family history of long QT syndrome.
22. Use or intend to use any prescription medications/products other than hormone replacement therapy, within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
23. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
24. Use or intend to use any nonprescription medications/products including vitamins, and minerals within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
25. Positive hepatitis panel. Subjects whose results are compatible with prior immunization may be included at the discretion of the Investigator.
26. Clinically significant abnormal laboratory values (clinical chemistry, hematology, coagulation, and urinalysis), as determined by the Investigator (or designee).
27. Significant history or clinical manifestation of hepatic disorder, as determined by the Investigator (or designee).
28. History or presence of liver disease or liver injury as indicated by any clinically significant deviations from normal reference ranges in liver function tests, unless approved by the Investigator (or designee).
29. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in (Day -1), or positive continine test at Screening or Check-in.

    For Subjects with Hepatic Impairment Only:
30. QTcF >450 ms (for mild and moderate hepatic impairment) or >470 ms (for severe hepatic impairment), confirmed by repeat measurement
31. Evidence of hepatorenal syndrome and/or estimated creatinine clearance range <90 mL/min (for mild and moderate hepatic impairment) or <60 mL/min (for severe hepatic impairment), as determined by the Investigator (or designee), calculated using the Cockcroft-Gault equation at Screening and Check-in (Day -1) For male subjects: ([1.23 × {140-age} × {weight in kg})])/(serum creatinine in μmol/L) For female subjects: ([1.04 × {140-age} × {weight in kg})])/(serum creatinine in μmol/L)
32. History of current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study including any of the following:

    1. Recent myocardial infarction (within 6 months of Check-in)
    2. New York Heart Association Class III or IV congestive heart failure
    3. Unstable angina (within 6 months of Check-in)
    4. Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, second or third degree atrioventricular block without a pacemaker
    5. Uncontrolled hypertension
    6. Unexplained syncope
33. Use or intend to use any prescription medications/products within 14 days of study drug administration, with the exception of stable medication regimen, as approved by the Investigator (or designee), Sponsor, and Covance Medical Monitor; see Inclusion Criterion #12; and prescribed hormone replacement therapy
34. Values outside the normal range for liver function tests that are not consistent with their hepatic condition, as determined by the Investigator (or designee).
35. Clinically significant abnormal PE, vital signs, and/or ECG findings that are not consistent with their degree of hepatic dysfunction, as determined by the Investigator (or designee).
36. Recent history, or the treatment of, esophageal bleeding (within the past 180 days of Screening), unless banded. If banded, it must not have occurred within 90 days of Screening.
37. Presence of a portosystemic shunt.
38. Recent history of paracentesis within 30 days prior to Check-in (Day -1).
39. Current functioning organ transplant or awaiting organ transplant.
40. Evidence of severe ascites.
41. Current symptoms or recent history of hepatic encephalopathy (Grade 2 or above) within 3 months prior to Screening.
42. Smoke more than 10 cigarettes, or use the equivalent tobacco- or nicotine-containing products, per day or inability to refrain from tobacco use 2 hours pre-dose until 4 hours post-dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
PK: AUC(0-inf) | Day 1 through Day 3
  Area under the concentration-time curve from time 0 to infinity
PK: AUC(0-t) | Day 1 through Day 3
  Area under the concentration-time curve from time 0 to the last measurable concentration
PK: C(max) | Day 1 through Day 3
  Maximum observed concentration
PK: t(max) | Day 1 through Day 3
  Time of the observed maximum concentration
PK: t(1/2) | Day 1 through Day 3
  Terminal elimination half-life
PK: t(last) | Day 1 through Day 3
  Time of the last measurable concentration
PK: CL/F | Day 1 through Day 3
  Apparent total clearance
PK: Vz/F | Day 1 through Day 3
  Apparent volume of distribution

SECONDARY OUTCOMES:
Safety: Incidence and Severity of Adverse Events (AEs) | Screening through Follow-up on Day 10
  Recording of the incidence, severity, relationship to KD025 of AEs and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Inland Empire Clinical Trials, LLC-HQ, Rialto, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Omega Research Group, Orlando, Florida
  - The Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Note: Undecided is not acceptable